CLINICAL TRIAL: NCT00133094
Title: Management of Hypercholesterolemia Utilizing a Case Management System, Incorporating Computer-Based Decision Support Technology
Brief Title: Systematic Management of High Cholesterol Utilizing Computer Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XVA 72-029; 00262
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-12

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Decision Support Systems, Clinical
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Simvastin; Procedure: Computer-based decision support technology

INTERVENTIONS:
Drug: Simvastin
Procedure: Computer-based decision support technology

SUMMARY:
Employing a physician-directed case management system, utilizing a Certified Registered Nurse Practitioner (CRNP) in conjunction with computer-based decision support technology (CDST) will result in significantly lower total cholesterol and a lower low density lipoprotein cholesterol in a group of subjects enrolled in a general medical clinic compared to subjects managed by primary care providers in the usual care group.

DETAILED DESCRIPTION:
Atherosclerosis affects 7 million patients and causes approximately 50% of all deaths in the United States. A reduction in modifiable risk factors (especially smoking, hypertension and hypercholesterolemia) is associated with a 30% reduction in acute coronary events. Clinically, fewer than 25% of patients achieve this degree of risk reduction because of significant barriers to implementation of effective risk reduction programs and wide variance in the management of hypercholesterolemia.

Recognition that a physician-directed case management system utilizing a certified registered nurse practitioner (CRNP) and computer-based decision support technology (CDST) offers the potential to implement disease management guidelines consistently and effectively is the impetus for this project. This project will demonstrate that enhanced compliance with the National Cholesterol Education Program (NCEP) guidelines can be achieved in a randomized trial conducted in subjects enrolled in a general medical clinic. The way in which hyperlipidemia will be managed is determined by randomization of the PCP providers to either the usual care group or to the intervention group, in which the management of subjects is delegated to the CRNP in conjunction with the CDST, under the supervision of the physician- investigators. Approximately 220 hypercholesterolemic subjects who are eligible for risk reduction according to NCEP guidelines will be recruited in equal numbers from subjects enrolled in the primary care clinic, beginning in 2005.

The physician-directed case management system employed in this project utilizes a management algorithm for lowering LDL-C cholesterol to the goal of less than 70 mg%. Stepwise increases in simvastatin dose to a maximum of 80 mg/day are used. Surveillance of symptoms and laboratory data to detect adverse side effects of the intervention precedes each increase in simvastatin dose. The CRNP will implement the management algorithm and concentrate on subject adherence, which is judged to be an important element in promoting compliance. The CRNP will initiate contact with the subject whenever a decision point is reached in the treatment algorithm, a deviation from the management algorithm occurs or an adverse reaction is detected. The case management model has been shown to be effective in achieving treatment goals in conditions such as hypercholesterolemia and diabetes mellitus.

This study will test hypothesis I, that employing a physician-directed case management system, utilizing a Certified Registered Nurse Practitioner (CRNP) in conjunction with computer-based decision support technology (CDST) will result in significantly lower total cholesterol and a lower low density lipoprotein cholesterol in a group of subjects enrolled in a general medical clinic compared to subjects managed by primary care providers in the usual care group.

A secondary aim of the project is to establish that computer-based decision support technology can be developed that will provide reliable clinical recommendations for the management of type II hyperlipidemia. This proposition will be tested by hypothesis II, that the computer-based decision technology provides advice for management of hyperlipidemia that is comparable to that of a cardiologist in the same institution.

Our physician-directed case-management system is expected to enhance guideline compliance by CDST monitoring of the subject�s compliance and cholesterol response to the management algorithm, thus contributing to improved outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of atherosclerosis and/or diabetes mellitus
2. Males age 45-70
3. Females age 55-70, at least 1 year post-menopausal
4. No contraindication to HMG-Co A inhibitor therapy
5. No administration of lipid lowering agents, except simvistatin less than or equal to 10 mg/day
6. TSH level greater than 0.34 and less than 5.6 IU
7. Urine protein less than or equal to 300 mg%
8. Lipid profile consistent with Fredrickson type hyperlipidemia: total cholesterol greater than or equal to 140 mg% and less than or equal to 300 mg%; LDL-C greater than or equal to 100 mg%; and triglycerides less than 400 mg%
9. Normal liver function tests (SGOT < 42 IU; SGPT <60 IU and CPK <269 IU)
10. One of the following diagnoses which establishes the presence atherosclerosis, making the subjects candidates for secondary prevention of complications or the presence of diabetes mellitus, which is considered an atherosclerotic equivalent according to the NECP III guidelines: uncomplicated acute myocardial infarction, more than 6 weeks previously; coronary arteriosclerosis (native artery and bypass grafts); prior aortocoronary bypass; prior PTCA; angina pectoris; peripheral vascular disease; or diabetes mellitus

Exclusion Criteria:

1) Women of childbearing age (2) Chronic liver disease and cirrhosis (3) Viral hepatitis, with residual hepatic dysfunction (4) Active alcohol abuse or dependence within the preceding 3 years (5) Drug abuse with or with out dependence within the preceding 3 years (6) Malignant neoplasms (7) Stroke (8) Dementia (9) Parkinson�s Disease (10) Multiple sclerosis (11) Triglycerides greater than or equal to 400 mg% (12) Other contra-indication to HMG-Co A administration such as cocomitant administration of drugs with known adverse interactions with simvastatin such as amiodarone, cimetidine, cyclosporin, tacrolimus, fibrates, HIV protease inhibitors, nefazodone, erythromycin, telithromycin clarithromycin, verpramil, itraconazole, ketoconozole, fluconazole danazol, or large quantities of grapefruit juice greater than 1 qt/day (13) Concurrent administration of lipid lowering agents or simvastatin at a dose greater than 10 mg/day at the time of entry into the protocol (14) Hypertension with systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg with or without treatment (15) Any chronic illness in which the life expectancy is <3 years such as oxygen-dependent COPD

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2006-06; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Total cholesterol and LDL-C cholesterol lowering

SECONDARY OUTCOMES:
Verification that the decision support program provides equivalent recommendations for management of elevated cholesterol as would an expert in the management of hypercholesterolemia

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ewing Thompson, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Click here for more information about this study: Management of Hypercholesterolemia Utilizing a Case Management System, Incorporating Computer-Based Decision Support Technology — http://www.cherp.org